CLINICAL TRIAL: NCT02956239
Title: Development, Field Testing and Evaluation of the Efficacy of a Hand-held, Portable and Affordable Thermo-coagulator to Prevent Cervical Cancer in Low- and Middle-income Countries
Acronym: DELTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: University of North Carolina Global Project Zambia (Unknown); Liger Medical Llc (Unknown)
Responsible Party: Principal Investigator, Partha Basu, Early Detection, Prevention and Infection Branch at IARC, WHO, International Agency for Research on Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1UH2CA202721-01 (NIH)
Record Dates: First submitted 2016-09-06; First posted 2016-11-07 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Cervical Precancer
Keywords: cervical precancer; screening; treatment; thermo-coagulation; thermal ablation; Reducing overtreatment
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Electrocoagulation; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thermocoagulation (device) (Experimental): VIA Positive women will be treated by the new device for thermocoagulation
  Interventions: Procedure: Thermocoagulation (device)
- Cryotherapy (device) (Active Comparator): VIA positive women will be treated by cryotherapy
  Interventions: Procedure: Cryotherapy (device)
- LEEP (device) (Active Comparator): VIA Positive women not suitable for thermo-coagulation or cryotherapy will be treated by LEEP
  Interventions: Procedure: LEEP (device)

INTERVENTIONS:
Procedure: Thermocoagulation (device) — Thermocoagulation uses heat injury to destroy the abnormal dysplastic cells of the cervix
  Arms: Thermocoagulation (device)
Procedure: Cryotherapy (device) — Cryotherapy uses cold injury to destroy the abnormal dysplastic cells of the cervix
  Arms: Cryotherapy (device)
Procedure: LEEP (device) — The abnormal area of the cervix is excised with a thin metallic loop driven by electrosurgical unit
  Arms: LEEP (device)

SUMMARY:
This project develops, tests and produces a lightweight, cordless, battery driven and rechargeable hand-held device for treating cervical precancer (Liger Thermal Coagulator). The study evaluates its effectiveness compared to the current standard treatment (cryocautery) when used as part of a screen and treat programme using Visual Inspection with Acetic acid (VIA) in Sub Saharan Africa.

DETAILED DESCRIPTION:
This project aims to improve screen and treat programmes for cervical cancers by discovering the best method of treatment. The specific aims are

1. To develop, test and produce 20 novel lightweight hand-held cordless, portable battery driven and rechargeable Thermal Coagulators (Liger Medical, Utah).
2. To evaluate the success / failure rate of Thermal Coagulation in a randomised controlled trial comparing thermal coagulation to the existing current standard cryocautery and to Large Loop Excision of the Transformation Zone (LLETZ aka LEEP) as part of a screen and treat programme in Zambia.
3. To evaluate the user satisfaction scores of the Liger Thermal Coagulator cryocautery as part of a screen and treat programme in Zambia.
4. To determine the rate of over treatment of VIA positive women as revealed by histopathological examination of the randomly assigned excised treatment cases.
5. To determine the value of Z scan to predict normality and abnormality in VIA positive women randomly assigned to excisional therapy

In collaboration with a medical devices company in Utah, the engineering performance of the Liger Thermal Coagulator has been developed and tested in vitro and in vivo. 200+ Liger units have been produced and a randomised controlled trial of the device has been undertaken, compared to cryocautery and LLETZ using efficacy and user friendliness as endpoints. The inclusion of a study arm of excisional therapy allows to quantify the rate of overtreatment in VIA programmes and using the Z scan may allow for a non invasive method of accurately predicting normality and abnormality in VIA positive women.

ELIGIBILITY:
Inclusion Criteria:

* Positive on VIA test for cervical cancer screening
* Eligible for ablative treatment

Exclusion Criteria:

* Pregnancy
* Not voluntarily willing to participate

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3124 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Difference in proportions with no lesions at 12 months follow-up between the thermocoagulation and cryotherapy arms among VIA positive women treated at baseline | 12 months
  The VIA positive women will be followed up after 12 months to see if the lesions have disappeared. HPV test will be used as the test of cure

SECONDARY OUTCOMES:
Over-treatment defined as the number of VIA positive women found with no CIN lesions in the post-operative LEEP specimens | 12 months
  The LEEP specimens will be subjected to histopathology to check for presence of cervical intraepithelial neoplasias

CONTACTS AND LOCATIONS:
Overall Officials: Partha Basu, Dr, Principal Investigator — IARC
Locations (1):
- UNC Global Project Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Pinder LF, Parham GP, Basu P, Muwonge R, Lucas E, Nyambe N, Sauvaget C, Mwanahamuntu MH, Sankaranarayanan R, Prendiville W. Thermal ablation versus cryotherapy or loop excision to treat women positive for cervical precancer on visual inspection with acetic acid test: pilot phase of a randomised controlled trial. Lancet Oncol. 2020 Jan;21(1):175-184. doi: 10.1016/S1470-2045(19)30635-7. Epub 2019 Nov 14. PMID 31734069
- [Background] Mwanahamuntu M, Kapambwe S, Pinder LF, Matambo J, Chirwa S, Chisele S, Basu P, Prendiville W, Sankaranarayanan R, Parham GP. The use of thermal ablation in diverse cervical cancer "screen-and-treat" service platforms in Zambia. Int J Gynaecol Obstet. 2022 Apr;157(1):85-89. doi: 10.1002/ijgo.13808. Epub 2021 Jul 31. PMID 34197624
- [Background] Basu P, Mwanahamuntu M, Pinder LF, Muwonge R, Lucas E, Nyambe N, Chisele S, Shibemba AL, Sauvaget C, Sankaranarayanan R, Prendiville W, Parham GP. A portable thermal ablation device for cervical cancer prevention in a screen-and-treat setting: a randomized, noninferiority trial. Nat Med. 2024 Sep;30(9):2596-2604. doi: 10.1038/s41591-024-03080-w. Epub 2024 Jun 25. PMID 38918630